CLINICAL TRIAL: NCT03576430
Title: The SongDance Study: Stress, Ongoing Self- Monitoring and Diabetes, Nerve Stimulation and Cognitive Empowerment
Acronym: SongDance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jens Faber, professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-17034836
Record Dates: First submitted 2018-05-22; First posted 2018-07-03 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2, Stress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: RCT, 1:1 inclusion active:control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active (Active Comparator): active stress handling
  Interventions: Device: active stress handling
- control (No Intervention): no stress handling

INTERVENTIONS:
Device: active stress handling — biofeed back stress handling
  Arms: active

SUMMARY:
Type 2 diabetes (DM2) I may be associated with low level of Quality of Life (QOL), depression, persistent stress and autonomic nervous system dysfunction (ANSD). A new biological measure measuring the Pressure Pain Sensitivity (PPS) of the chest bone has been found to be a marker for persistent stress and ANS function, and linked to depression, QOL, chronic inflammation and HbA1c. An intervention which uses the PPS measure as a biological feedback marker for stress reduces the level of persistent stress (PPS) and depression, reduces blood pressure, serum lipids, restores ANSD and increases quality of life.

Objectives: primary: if a simple individualized self-care based intervention, using the PPS of the chest bone as a biofeedback marker for stress, reduces PPS and with concomitant reduction in HbA1c. Secondly, if changes in PPS and HbA1c correlate, if the level of depression and number of clinical stress symptoms are reduced, and QOL and personal empowerment increased. Thirdly, if use of glucose-lowering medication, blood pressure, heart rate, work of the heart, autonomic nervous system dysfunction measured by PPS and cardiovascular response to tilt table test and heart rate variability, serum lipids and low-grade inflammation are reduced. As a separate part of the study, the implementation aspects of the PPS guided intervention are studied.

Design:RCT,single-blinded, 1:1 randomization, in which diabetic treatment as usual (TAU) is compared to TAU plus a self-care based intervention program based on daily PPS measurements at home over a 6 months period and daily 2 times nervestimulation as mandatory. The study will be open to the patient and the treating professionals but blinded towards the evaluating researchers. The implementation part of the study will be conducted according to WHO guidelines.

Patients: 160 patients with DM2 from primary health care. Effect variables: Primary: HbA1c. Secondary : PPS, depression, QOL, personal empowerment, and the correlation between changes in PPS and HbA1c.

Treatment: All patients receive diabetes care as usual. The active group receives in addition the self-care based, non-pharmacological PPS guided intervention program, which focuses on daily PPS measurement for cognitive reflection and cutaneous sensory nerve stimulation for reduction of PPS with the aim to reduce the elevated PPS.

DETAILED DESCRIPTION:
Introduction About 350 million people worldwide have type 2 diabetes (DM2). Approximately 85% of these patients are controlled in the primary health care.

A high level of personal care, i.e. high empowerment, is a pre-requisite for successful outcome of their diabetes disease. Therefore, all patients are encouraged to measure their blood glucose levels several times a week or daily, depending on the type of treatment, and to act according to the blood glucose level, typically by changing lifestyle. Several studies have shown that high empowerment increases QOL in diabetes patients. In general, living with a chronic disease is associated with low QOL, fear of the future, anxiety and depression, and similarly for patients with DM2. These elements may lead to a state of chronic stress.

The link between persistent stress on the one side, and chronic arterial inflammation and cardiovascular events recently received support from a long-term study using region brain activity as assessment for chronic stress

The PPS measure and the PPS-guided intervention Persistent stress or allostatic overload as it is also called can be measured using an algometer measuring the pressure pain sensitivity at the sternum (PPS), and the measure can be used as self-monitoring at home using daily measurements. This can then be followed by action, and thus increase the personal empowerment.

In an intervention study in healthy office workers, it was found that a reduction of an elevated PPS was significantly associated with a reduction in HbA1c, blood pressure, serum lipids, body mass index, serum YKL 40 (a marker of inflammation),and ANS dysfunction

In another chronic disease, ischemic heart disease, we have demonstrated that daily measurement of one's individual stress levels by this algometer followed by nerve stimulation as a mandatory stress modulating treatment (the ULLCARE program) reduced depressive symptoms, increased well-being and quality of life and restored ANSD The concept: measure PPS and take action aiming at reducing the persistent stress load in chronic disease is thus established.

In a pilot study (n=100), approximately 70% of DM2 patients had an elevated PPS measure (≥ 60), indicative of presence of persistent stress.

The guidelines of WHO for implementation research will be applied in the present study

Rationale of the study The pharmaceutical treatment in DM2 is associated with potential side effects, is associated with health care expenses and may in the long run show to be insufficient to keep blood glucose low.

On this background, the search for non-pharmaceutical selfcare-based interventional modalities that increase patient empowerment become attractive. The present intervention represents one such intervention. Further, application of the concept to the most vulnerable patients with ischemic heart disease has an effect size on depression much larger than anti-depressive medication.).

Hypothesis A simple individualized self-care based intervention program, that uses frequently PPS measure as a feedback marker of stress followed by cutaneous sensory nerve stimulation, reduces the level of persistent stress measured as PPS, and concomitantly reduces HBA1c, depression, clinical stress score, and increase QOL and empowerment, and by this reduces the use of glucose-lowering medication.

Research questions

Does the self-cared based intervention program ULLCARE, with focus on PPS measurement as biofeedback marker of stress and nerve stimulation as mandatory plus free-of-choice own efforts for stress reduction, help patients with DM2 through increased self-care over a six months period leading to:

Reduced persistent stress measured as PPS Reduction of an elevated HbA1c Reduction in depression and clinical stress score, and improved QOL and empowerment Correlation between reduction in PPS and reduction in HbA1c among patients with HbA1c ≥ 53 mmol/mol at baseline, PPS ≥ 60 arbitrary units at baseline, and who obtain a reduction in PPS ≥ 15 arbitrary units during intervention period Reduction in use of glucose-lowering medication Reduction in blood pressure, heart rate, work of the heart, low grade inflammation (i.e. YKL 40), ANS dysfunction, serum lipids, BMI and visceral fat

Implementation research questions:

As a separate part of the study, the implementation aspect of the PPS guided intervention is as studied according to the WHO implementation study guidelines:

Questions at 6 months follow-up up

Patient evaluation of the intervention program: Among others:

How long did it take you to become familiar with the use of the PPS measurement device? To what extend do have you found the use of the PPS measurement device useful? Does the PPS measure serve its purpose, to increase sense of increased personal control? Are the mandatory daily PPS measurement and nerve stimulation acceptable and feasible?

Design A prospective, randomized observer-blinded controlled trial in which the effect of a 6 and 12 months PPS guided selfcare based intervention program plus treatment as usual (TAU) (e.g. active group) is compared to a control group, who receives TAU.

Blinding and randomization The study is open to the participating patients and the instructors of the active group. The study is blinded to all others, including the statisticians who make the main analysis. The personnel conducting the clinical examinations does not have access to the documents containing information about the treatment or treatment procedures. This is to prevent bias in the comparison between the treatment groups.

The study endocrinologist, who regulates all glucose-lowering, lipid-lowering and blood pressure-lowering medication, is blinded to the group allocation.

Randomization is 1:1, active: control. An independent research company electronically conducts the practical randomization. The result of the randomization is blinded to the investigating personel besides the people conducting the training of the active group as well as patients are excluded from blinding.

The patients are stratified in three groups: HbA1c below 53 mmol/mol: HbA1c: 53 - 63 mmol/mol; HbA1c: 64 - 75 mmol/mol.

Material 160 patients recruited from primary health care will be included.

Further, the first 50 patients who meet the inclusion and exclusion criteria in all aspect, except by having a PPS value below 60, will be invited to participate in the full baseline examination.

Inclusion criteria: see elsewhere Exclusion criteria : see elsewhere Outcome measures : see elsewhere Previous studies have shown that when an elevated PPS is reduced, the secondary effect on other outcome measures is larger, if these outcome measures are elevated at baseline as well

On this background, the present study will focus on effect on these outcome measures, when they are elevated at baseline. Discrimination values for each outcome measure will be as follows:

HbA1c: ≥ 53 mmol/mol PPS: ≥ 60 arbitrary units Blood pressure: ≥ 130/85 mm Hg Heart rate: ≥ 70 beats/minute Depression score; MDI ≥ 15 WHO 5: score < 50 arbitrary units Clinical stress score: ≥8 arbitrary units Total cholesterol: ≥5.0 mmol/L LDL cholesterol: ≥3.5 mmol/L HDL cholesterol: ≤ 0.9 mmol/L Triglyceride: ≥ 2.0 mmol/L

Implementation related outcome measures:

User feedback addressing the:

educational program, conduction of the program at home, the professional support and the web related support.

Provider feedback among the professional staff taking care of education and professional support

Use of glucose-lowering medication The treatment target for glycemic control is 48 mmol/mol. Reduction in HbA1c to a level above or equal to 48 mmol/mol does not lead to change in medication In patients with a HbA1c below 48 mmol/mol a further reduction of 3 mmol/mol will lead to an evaluation with respect to reduction in anti-diabetes medication performed by the study diabetologist, blinded to the randomization and according to Danish National Guidelines If the patient experiences a hypoglycemic episode, she or he is asked to contact the study nurse, and the study diabetologist will consider whether change in glucose-lowering medication is needed.

If HbA1c increases more than 3 mmol/mol at any point at follow- up, the glucose lowering medication is evaluated with respect to an increase in anti-diabetic medication and according to the judgement of the study diabetologist and according to Danish National Guidelines. The study diabetologist is blinded to the randomization.

Intervention Control/Active group:

Control group: continue their diabetes care program as usual

Active group: receive in addition to the above mentioned:

Instruction in UllCare program during a 45 minute personal consultation by a UllCare program instructor certified nurse Mandatory daily efforts: Self-measurement of PPS to be done twice daily; Nerve stimulation according to instruction; Use of personal web journal Free-of-choice modalities for further reduction of the PPS measure if needed. The patient receives the following instruction material: An Ull Meter, a written instrument instruction manual, a booklet with the Ull Care intervention program, a DVD instructor manual for use of PPS measurement device and nerve stimulation, and a log-in for their personal web journal Five telephone consultation with the UllCare instructor after 1,3, 5, 6 and 10 weeks Two face-to-face consultations with UllCare Instructor at 1 and 3 months The patients record their PPS measurements either on a web platform or on paper at least once a week If their PPS records show a PPS ≥ 60 for 7 consecutive morning measurements, the patient is contacted regarding the need for additional technical instruction.

After six months of participation in the project all patients (both groups) are called to a repetition of the baseline visit at Herlev Hospital.

The two examinations at Herlev hospital are conducted by the same blinded nurse at baseline and the 6-month follow-up respectively.

Data with respect to the outcome measures of the study may also be obtained from the patient record at www.sundhed.dk After 12 months data with respect to HbA1c and use of glucose-lowering medication is obtained through the public data.

In case blood glucose/HbA1c increases In this case the diabetologist, which is blinded to the treatment allocation, will decide which potential changes in medication should be done. In case the General Practitioner wants to change blood pressure medication or lipid lowering medication, he or she is urged to inform the study nurse.

Methods PPS measurement An Ull Meter is used, which is an instrument developed to measure the sensibility/activity in the polymodal nervous system corresponding to the most painful point on the sternum between costa 3-5. The point is identified by finger pressure. First the patient learns his/hers pain threshold as the instructor applies a gradually increasing pressure on the distal phalanges of the left index finger with the instrument and the patient is instructed to say stop when the threshold of pain/discomfort is reached. If the instructor observes a withdrawal reflex (i.e. an involuntary muscle contraction of the muscles around the eyes, the neck or upper limb) before the patient says stop, the procedure is stopped as well. The procedure is then repeated on the most tender place on the sternum. The instrument then displays a number on a scale from 30 to 100, where an increased sensibility is accompanied by an increasing number, PPS; meaning that a high PPS measure reflects a high level of stress (high sensitivity). The PPS is determined as the average of two consecutive measurements on the same location on the sternum and with 5 seconds between measurements. If difference between the two measurements exceeds 10 PPS arbitrary units, a third measurement is conducted and the average between the three measurement is used as the PPS measure.

The Ull Meter has the following special features:

Hidden measurement value until the measurement is completed. A calculation of the sensitivity to a tenderness score on a logarithmic scale similar to the decibel scale used to estimate the limit values of sound pressure in connection with a hearing test.

An alarm that is activated by a pressure before the occurrence of any injury. A special foot pad that prevents irritation of the skin to ensure that it is the pressure sensitivity of the bone that is measured and not the skin's sensitivity.

Treatment modalities

Current diabetes care:

At baseline, all patients received standard diabetes care according to national guidelines, which include medical counselling by the study nurse, medical standardization by the study diabetologist, education in DM2 and life style adjustments.

The Ull Care program:

The basic elements of the intervention are as follows:

A self-care part. A professional instruction in the PPS measurement, cognitive reflection in relation to the measure and nerve stimulation.

Continuous recording of the participants' PPS measurements through a Web journal.

The self-care based intervention program is a stress management program based on the use of the PPS measure as a biofeedback marker of stress. The most important effort is the daily self-care in the form of PPS measuring, cognitive reflection and nerve stimulation, which is linked to professional technical help depending on need.

The elements of the self-care program An individual start-up of a 45-minutes face-to-face consultation at home with an Ull Care instructor who explains the use of the instrument, the interpretation of the PPS measurement, nerve stimulation and the web platform.

A personal Ull Meter instrument. A personal web journal for track recording of the participant's PPS measure's development (patients without internet access will receive printed registration sheets).

A booklet that describes the self-care program in details. Two additional face-to-face meetings with additional professional instruction should the PPS measure remain ≥ 60 after 1 and 3 months respectively.

5 x 15 minutes of telephone consultations after 1, 3, 5, 6 and 10 weeks respectively.

Online assessment of the participant's PPS measurements. This assessment is made automatically on the website.

Professional support: If the morning PPS measure has been ≥ 60 for more than seven days in a row, the participant is contacted pro-actively and offered additional professional support with the overall aim in mind: obtain and main low PPS measure, preferable < 45, and acceptable < 60 arbitrary units.

The daily steps of the self-care program Four elements constitute the daily self-care system: measuring, cognitive reflection, action and control.

Measuring: PPS is measured twice a day as a fully private measure and is entered in a personal web journal, so that the person can track his/hers own development, while at the same time there is a regular external professional control.

Reflection: Cognitive reflection as a reaction to the actual PPS measure and its development. Action: Nerve stimulation on selected acupuncture points corresponding to the instruction. Possible further own efforts are as mentioned in the book on general stress management given to all participants (both the active and control group). The PPS measure is used as a personal feedback marker of stress, taking into account the effect of the participant's chosen effort.

Control: Measure the effect of any action/inaction at any time.

This four-step procedure should be done at least twice a day (morning and evening) to be preventive; it is recommended to perform the procedure morning and evening in order to promote the construction of a conditioned reflex. This reflex (i) facilitates the habit and (ii) improves the effect of the action, which is important for ad-hoc use, should the participant want to reduce his/hers level of stress acutely or if he/she experience one or more of the clinical stress symptoms, which is presented to her/him as part of the educational program.

The specific therapeutic elements of the program:

Daily mandatory efforts Biofeedback measuring of stress using the PPS measure as composite measure for important diabetes risk factors which are possible to influence by the suggested own efforts.

Sensory nerve stimulation (acupressure/shiatsu massage) Free-of-choice supplementary own efforts. As the main effort of the program is to reduce an elevated PPS measure, additional own-efforts will be recommended on an individual basis in response to the observed reduction in PPS or lack of such reductions. Such efforts included a variety of physical, mental, emotional, social modalities as well as diet recommendations. These modalities are presented to the patient as part of the written educational material

PPS measurement

The patients are instructed to perform the PPS measurement twice daily, similarly and as a supplement to the home blood sugar measurement. It is explained that:

the PPS measure represent a simple and reliable composite measure for a variety of important diabetes and cardiovascular health risk factors, including HbA1c, autonomic function, blood pressure, heart rate, work of the heart, serum lipids, low grade inflammation, QOL, depression and persistent stress.

That all of these risk factors improves concomitantly (if elevated) when PPS is persistently reduced to a level below 60 arbitrary units and with the ultimate goal to obtain a morning PPS below 45 arbitrary units.

That the present PPS guided self-care based non-pharmacological intervention will do the job when applied on a daily basis, similarly to the daily tooth brushing for caries prevention.

Nerve stimulation:

The patients are instructed to perform the preventive nerve stimulation twice a day plus ad hoc when they urgently want to reduce their stress. Nerve stimulation is done by applying pressure with a finger for one minute - you should feel it, but it should not cause any pain, This is done at the following acupuncture points; on the sternum at the level of the fourth intercostals space (Shanzhong, C.V. 17), and on the back 3,8 cm lateral to the spinal process of the fourth and fifth thoracic vertebra (Jueyinshu and Xinshu, U.B. 14 and 15) Nerve stimulation is done successfully when the patient can observe that the tenderness of the point has been reduced after applying pressure for 20 to max 60 seconds. If this result has not been achieved, the patient is instructed to repeat the treatment. The repetitive nerve stimulation has two primary goals: 1) to restore the nervous system's ability to adapt through the repetitive stimulation of the diffuse pain inhibitory control (DNIC) system and 2) to reduce an elevated stress level through the repeated non-painful sensory stimulation of the polymodal nerve cell, causing a release of the oxytocin hormone. If possible, the spouse or cohabitant will be instructed to perform nerve stimulation on the patient's back, which may independently contribute to stress-relieving effects through a separate oxytocin release caused by the human care. If a spouse or cohabitant is not available, the patient can perform the treatment himself with a ball (the person will receive instructions in the technique).

Blood analyses Blood samples are taken locally at Medical Department , Endocrinology Unit, Herlev Hospital. Routine analyses as HbA1c is measured immediately at. After analysis, and by June 1st 2021, the debris is destroyed.

Besides this a blood sample is taken and stored at -80 degrees until analysis. This is for research purpose. All research analysis will performed at Medical Department , Endocrinology Unit, Herlev Hospital. All samples are analysed in the same assay to avoid inter-assay variation, i.e. the analyses are first performed after completion of the study.

Besides this, a spare sample of 20 ml of blood is taken for any later use at baseline and at the 6 months follow-up. These spare sample are stored in coded form (without CPR number) in one of the Danish Data Protection Agency and the Capital Region's approved bio banks (database id: 30122009.HEH.O.JF). This database is an ongoing database without a planned end date. The aim of this data bank in supplementary blood analyses for research purpose.

Questionnaires

The following questionnaires will be included as outcome measures:

1. Diabetes empowerment is measured by the questionnaire DES-SF
2. Major depression inventory (MDI)
3. WHO-5 quality of life score
4. Clinical stress sign score
5. SF-36 for physical and mental health
6. Epworth Sleepiness score
7. Diabetes treatment satisfaction questionnaire

other measures BMI: will be measured as weight in kilogram divided with height in meters squared.

Blood Pressure (mm Hg) and pulse (beasts/minute: measured automatically conducted in the supine position after 10 minutes of rest Work of the heart is measured as Pressure-Rate-Product (mm Hg/beats per minute: systolic blood pressure x heart rate Body Composition (visceral fat): measured by Omron BF 500, 4-point bio electrical impedance measure, using metal footpads and hand electrodes

ANS measure:

* HRV measured by Vagus instrument (non-invasive procedure)
* Table tilt testing: standardized procedure tilting the subject to 70 degrees and measure blood pressure, pulse rate and PPS before and after 7 min tilting

Statistics Calculation of sample size and power analysis Calculation of sample size is based on the followed premises with respect to HbA1c. The Minimal Important Difference is 4 mmol/mol; mean HbA1c as baseline is estimated to be 64 mmol/mol, and with standard deviation: 9 mmol/mol. Alfa: 5%, Beta: 80 %. This lead to 160 as total sample size.

The Minimal Important Difference with respect to effect size is calculated as per protocol (i.e. all patients who complete the study, including the 6 months follow-up examination) as well as on all included patients on intention to treat basis. .

Cohens effect size is a fraction that consists of the difference in a HbA1c from before intervention till after treatment for the active group, minus the same difference for the control group divided by the spread (i.e. standard deviation) of the change in HbA1c, when taking all patients together. Example: the HbA1c in active group changes from 64 to 56 (64-56) = 8 mmol/mol; while the HbA1c for the control group changes from 64 to 60 (64-60) = 4 mmol/mol. This change in the HbA1c is 8-4 = 4; if the spread on the HbA1c for all patients is 9, the effect size will be 4/9 = 0.4.

Analysis of the effect variables Five percent (5 %) will be used as significance level in all statistic tests. The statistics are compiled on an "per protocol" and "intention to treat basis". The former meaning that all patients who complete the trial are included; the latter meaning that all enrolled patients are included in the subsequent analysis. Both set of analyses will be published.

Delta values (i.e. difference between baseline and follow-up measurement) for the active and control group respectively will be compared to analyse for a possible treatment effect. All secondary and tertiary effect variables will be analysed after the intervention through variance and regression analysis. If the premises for the proposed statistical analysis cannot be met, non-parametric analysis is used. Quality-of-life data will be analysed to meet the directions of each of the questionnaires. All effect data will be presented a unifying table and primary, secondary and tertiary effect variables will be listed.

With respect to calculate the effect with respect to outcome measures, which are elevated at baseline, these will be calculated for the group of patients who has an elevated risk profile with respect to the individual outcome measure (e.g. when triglyceride is tested for change, this is done among the patients with an elevated triglyceride level at baseline). These effect variables include: triglyceride, Total cholesterol, HDL- and LDL cholesterol, blood pressure, heart rate and Pressure-Rate-Product, glycated hemoglobin, PPS, MDI depression score and WHO5 well-being score (see point 5: outcome measures). The proportion of patients who obtain such effect will be compared between the two groups of patients: those who experience a reduction of PPS ≥ 15 arbitrary units, and those who do not.

Glucose-lowering medication: it will be calculated as between-group differences in the proportion of participants who: (i) reduce the use of glucose-lowering medication, (ii) who totally discontinue the use, and (iii) who increase their use. The between-group difference in proportion of patients who reduce, discontinue or increase their use of glucose-lowering medication will be calculated using 2x2 Contingency table test

Success criteria The first priority criterium for a successful outcome of the study is a significant between group difference. Secondly, effect size calculated as described in Statistics section of this protocol

Benefits for the patients By participating in the study, each patient can get a general profit from the opportunity of an additional comprehensive health check. If the findings of the study are positive, it means that the patients in the active group have an extra benefit in terms of improved glycemic control, increased empowerment, reduced stress, improved QOL, reduced glucose-lowing medication and some concrete tools for maintaining these benefits

Ethics The study is approved by the local Scientific Ethics Committee. The study is also reported to the Danish Data Protection Agency. The study complies with the Helsinki Declaration.

All subjects are informed orally and in writing about the study. The subject's right not to receive information on his/hers health condition and disposition to disease will be reviewed and respected.

If the subject gives written permission, two spare blood sample will be stored from both baseline and the month follow-up in one of the Danish Data Protection Agency's approved bio banks (jr.nr 2005-41-5655, later 2008-41-2031, and from Dec 2009: 30122009.HEH.O.JF).

There will be no financial compensation to subjects. If during the conduct of the trial new information on effect, risks and side effects appear, the subjects will be informed, and a new informed consent may be obtained.

Use of the blood samples for any other purpose than what the subjects initially consented and what is referred to in this protocol will follow the usual guidelines, including a renewed reporting to the ethics committee.

Risks and rights and information of the participants The patients are not deprived of other known effective treatment, and participation in the study does not interfere with the patient's current treatment.

The patients will be asked for permission to take an extra blood sample for research purpose.

By measuring the pressure threshold, some soreness or bruises may occur if the participant does not follow the instructions.

The HRV position testing is non-invasive and without discomfort or risk to the person.

The given active intervention is risk-free.

The initial contact from the study group to the patient is by invitation presented in public media and to the local general practitioners. The first contact is a telephone call from the patient to the study nurse. Secondly, the patient come to Herlev Hospital for a personal information consult with the study nurse, and which takes place in a room with no other persons around. For this meeting, the patient is recommended to bring an assessor. Furthermore, at this consultation the patient receives the following documents 1) "Deltagerinformation, 2) "Samtykkeerklæring", 3) "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt", og 4) "før du beslutter dig". For this consult, there will be emphasis on the fact that the information session is about a query of participation. The subject's right not to receive information on his/hers health condition and disposition to disease will be reviewed and respected.

Thirdly, if the patient wants to participate, the "Samtykkeerklæring" must be returned to the study nurse, preferable within a week after the information consult. Thereafter, the patient is scheduled for baseline examination.

Conflicts of interest Søren Ballegaard is a shareholder in Ull Care A/S and is the inventor of the Ull Meter. To minimize possible bias, he shall not participate in 1) patient selection, and 2) evaluation of the treatment. Jens Faber, Finn Gyntelberg and Ebbe Eldrup do not own shares or other financial interests in Ull Care A/S and have never received funding/fees from the company. Thus they have nothing to declare as disclosures.

Wirth respect to the use of the DES-SF questionnaire, the project described was supported by Grant Number P30DK092926 (MCDTR) from the National Institute of Diabetes and Digestive and Kidney Diseases.

Substudy By the use of public registers (i.e. www.Sundhed.dk, it is the intention to conduct a 12 months follow-up with respect to 1) HbA1c and 2) use of glucose lowering medication. Secondly to record the implementation aspect of the study. Presently, financial support for this sub study is applied for.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

* Diagnosed DM2,
* HbA1c: ≤ 9 % (75 mmol/mol)
* BMI < 40.
* PPS ≥ 60 units;
* Age < 75 years;
* Manage the Danish language for proper use of instructions,
* Actively express to accept to conduct minimum 20 minutes of self-care daily.

Exclusion Criteria:

* Use of insulin as basal-bolus regime (i,.e. the combination of long-term acting insulin as basal insulin and short-term lasting insulin as bolus injections before meals)
* Use of Beta blockade medication
* HbA1c > 9 % (75 mmol/mol)
* Previously diagnosed and treated for a psychiatric disorder, except for depression.
* A chronic competing disorder that statistically is life-shortening (such as advanced cancer with metastases).
* A chronic competing disorder that is not heart disease and which clearly impairs the patient's quality of life /e.g. COPD, cancer, chronic pain syndrome).
* Patients who cannot fend for themselves.
* One or more of the following complications: diabetic retinopathy that needs specific treatment, or nephropathy (i.e. plasma creatinine ≥ 200 umol/L))

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C | 0, 3 and 6 months
  numeric scale 30-150 mmol/mol; higher value indicates worsening of diabetes control

SECONDARY OUTCOMES:
pressure pain sensitivity | 0, and 6 months
  numeric scale, range 30-100; higer values indicate more stressed person
Correlation between changes in pressure pain sensitivity and Hemoglobin A1C | 0, and 6 months
  see above, numeric scale; range 0-1, higher correlation indicates higher association between mean bood glucose and stress
Personal diabetes empowerment scale (DES-ST) | 0, and 6 months
  4 questions, range 1-5, sum score, numeric scale range 4-20; higher values indicate higher empowerment
quality of life index (WHO-5) | 0, and 6 months
  5 questions, sum score, numeric scale, range 0-25, higher values indicate better quality of life
Physical and mental health (SF 36) | 0, and 6 moths
  quality of life, 11 questions, sum score, numeric scale, range 0 - 100; higher values indicate better Physical and mental health
Depression (MDI questionnaire) | 0, and 6 moths
  depression symptoms, 10 questions, range 0-6, sum score, numeric scale, range 0-60; higher values indivate more depressed person
Number of clinical stress symptoms measured by a specially designed questionnaire | 0, and 6 moths
  Number of stress symptoms, sum of 56 questions, numeric scale; range 0-56, higher values indicate more stressed person
Sleepiness score (Epworth) | 0, and 6 months
  8 questions, range 0-3, sum score, numeric scale; range 24; higher values indicate increased tiredness
Diabetes treatment satisfaction questionnaire (DTSQ) | 0, and 6 months
  treatment satisfaction: 8 questions, range 0-6, sum score; range 0-48, the higher the more satisfied

OTHER OUTCOMES:
blood pressure | 0, and 6 months
  measured in mmHg, numeric scale with no min and max range; higher values indicate more stressed person
Autonomous nervous system function measured by Heart Rate Variability (HRV) and by the blood pressure, heart rate and PPS response to a Tilt Table test | 0, and 6 months
  HRV: measured by beat-to-beat variation during rest, numeric measure , range 0-3; the higher the value the more Autonomous nervous system dysfunction
Change of glucose-lowering medication | 0, 3 and 6 months
  medication is reduced at 3 and 6 months treatment based on an algoritm using change in Hemoglobin A1c from baseline as decision factor
table tilt testing, effect on Pressure pain sensitivity | 0, and 6 months
  autonomous nervous system testing: Pressure pain sensitivity is measured before and after tilting. Scale numeric; range 0-70; the higher value the better the autonomous nervous system
resting pulse rate | 0,and 6 months
  measured in beats/min; numeric scale, no min and max value; higher values indicate more stressed person

CONTACTS AND LOCATIONS:
Overall Officials: jens faber, professor, Principal Investigator — Herlev Hospital
Locations (1):
- Department of Medicine, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faber J, Eldrup E, Selmer C, Pichat C, Hecquet SK, Watt T, Kreiner S, Karpatschof B, Gyntelberg F, Ballegaard S, Gjedde A. Reduction of Pressure Pain Sensitivity as Novel Non-pharmacological Therapeutic Approach to Type 2 Diabetes: A Randomized Trial. Front Neurosci. 2021 Mar 11;15:613858. doi: 10.3389/fnins.2021.613858. eCollection 2021. PMID 33776633